CLINICAL TRIAL: NCT02719470
Title: Does Cognitive Impairment Affect Rehabilitation Outcome in Parkinson's Disease?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cognition and reahb in PD
Record Dates: First submitted 2016-03-06; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease
Keywords: Cognition Impairment; Rehabilitation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- normal cognition (Experimental): Group 1: patients with normal cognitive profile, assessed with MMSE (27 ≤ correct score ≤ 30) undergoing MIRT
  Interventions: Behavioral: MIRT
- mildly impaired cognition (Experimental): Group 3: patients with middle cognitive decline, assessed with MMSE (20 ≤ correct score < 27) undergoing MIRT
  Interventions: Behavioral: MIRT
- moderately-severely impaired cognition (Experimental): Group 2: patients cognitive decline, assessed with MMSE (correct score < 20) undergoing MIRT
  Interventions: Behavioral: MIRT
- patients with normal executive functions (Experimental): Group 4: patients with pathological executive functions, assessed with FAB (FAB ≥ 13.8) undergoing MIRT
  Interventions: Behavioral: MIRT
- pathological executive functions (Experimental): Group 5: patients with pathological executive functions, assessed with FAB (FAB < 13.8) undergoing MIRT
  Interventions: Behavioral: MIRT

INTERVENTIONS:
Behavioral: MIRT — MIRT consists of a 4-week physical therapy, in a hospital setting, which entails four daily sessions for five days and one hour of physical exercise on the sixth day. The duration of each session is about one hour. The first session consists of a one-to-one session with physical therapist involving muscle stretching. The second session includes aerobic exercises to improve balance and gait using different devices: a stabilometric platform, treadmill plus, crossover and cycloergometer. The third is a session of occupational therapy to improve autonomy in everyday activities. The last session includes one hour of speech therapy

SUMMARY:
In order to explore the question how an intensive, goal-based and aerobic rehabilitation treatment, addressed to act on motor and mental aspects, affects motor and functional symptoms in PD patients with normal cognition and with different level of cognitive impairment. Hypothesis is that a specific rehabilitation program based on motor-cognitive training and repetition, can affect positively the rehabilitation outcome regardless of baseline cognitive profile.

DETAILED DESCRIPTION:
Objective: This study is aimed to evaluate the impact of cognitive decline on rehabilitation outcomes in Parkinson's disease (PD). While cognitive status is considered as a determinant of rehabilitation outcome, no studies about this issue have been performed before.

Methods: 438 PD patients hospitalized for a 4-weeks Multidisciplinary Intensive Rehabilitation Treatment (MIRT) were enrolled. According to Mini Mental State Examination (MMSE), patients were divided into: normal cognition (MMSE 27-30), mild cognitive impairment (MMSE 21-26), moderate or severe cognitive impairment (MMSE ≤ 20). According to Frontal Assessment Battery (FAB), subjects were divided into patients with normal (FAB ≥ 13.8) and pathological (FAB < 13.8) score. The outcomes measures were: Unified Parkinson's Disease Rating Scale (UPDRS), Berg Balance Scale (BBS), Timed Up and Go Test (TUG), Six Minutes Walking Test (6MWT), Parkinson's Disease Disability Scale (PDDS).

ELIGIBILITY:
Inclusion Criteria:

* Parkinsonian patients according to the UK Brain Bank criteria

Exclusion Criteria:

* Major stroke, possible hydrocephalus or brain tumor observed on CT scan or brain MRI
* Major depression, active psychosis or clinically significant psychiatric disorders
* Visual or auditory disturbances that prevent the neuropsychological assessment
* The increase in drug dosage during hospitalization

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | 4 weeks

SECONDARY OUTCOMES:
Berg Balance Scale | 4 weeks

OTHER OUTCOMES:
Timed Up and Go Test | 4 weeks
Six Minutes Walking Test | 4 weeks
Parkinson's Disease Disability Scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital - Gravedona ed Uniti (CO, Italy)
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No